CLINICAL TRIAL: NCT07374757
Title: Clinical Outcomes of Immediately Loaded Implants With Buccal Dehiscence Treated by Horizontal Augmentation Compared With Immediately Loaded Implants Without Regeneration Techniques
Brief Title: Immediately Loaded Implants With or Without Horizontal Augmentation
Acronym: ILHA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCM2026
Record Dates: First submitted 2026-01-20; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Bone Augmentation Associated With Immediate Loading
Keywords: Inmediate loading; horizontal bone regeneration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Horizontal bone augmentation associate with immediate loading (Experimental): Horizontal bone augmentation associate with immediate loading
  Interventions: Procedure: guided bone regeneration technique
- Inmediate Loading without bone regeneration technique (Other): Immediately loaded dental implants placed without the use of any bone regeneration or augmentation techniques.
  Interventions: Procedure: No intervention

INTERVENTIONS:
Procedure: guided bone regeneration technique — Immediately loaded dental implants placed in sites presenting buccal dehiscence treated by horizontal bone augmentation using a guided bone regeneration technique according to a standardized surgical protocol.
  Arms: Horizontal bone augmentation associate with immediate loading
Procedure: No intervention — Immediately loaded dental implants placed without the use of any bone regeneration or augmentation techniques.
  Arms: Inmediate Loading without bone regeneration technique

SUMMARY:
This study aims to compare the clinical success and patient-reported outcomes of immediately loaded dental implants placed in sites with buccal dehiscence treated by horizontal augmentation versus immediately loaded implants placed without regeneration techniques.

DETAILED DESCRIPTION:
This is a prospective, interventional, non-randomized, comparative clinical trial designed to evaluate the clinical outcomes of immediately loaded dental implants using two different surgical approaches. One group will receive implants placed in sites with buccal dehiscence treated by horizontal bone augmentation, while the comparison group will receive immediately loaded implants placed without the use of any bone regeneration techniques.

The primary outcome of the study is implant success at 12 months after implant placement. Secondary outcomes include marginal bone level changes, complication rates, and oral health-related quality of life assessed using a validated questionnaire. The study is conducted with a parallel assignment model and an open-label design due to the nature of the surgical interventions.

ELIGIBILITY:
Inclusion Criteria:

Adult patients requiring dental implant placement Presence of buccal dehiscence at the implant site Indication for immediate loading Ability to provide written informed consent

Exclusion Criteria:

Uncontrolled systemic diseases Active periodontal disease Heavy smoking exceeding predefined limits Conditions contraindicating oral surgery

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-08 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12-11 (Estimated)

PRIMARY OUTCOMES:
Implant Success Rate | 12 months after implant placement
  Implant success is defined as implant survival at 12 months, absence of clinical mobility, absence of persistent pain or infection, absence of peri-implant radiolucency, and no need for implant removal or surgical re-intervention.

IPD SHARING:
Plan to Share IPD: Undecided